CLINICAL TRIAL: NCT04322344
Title: Efficacy and Safety of Escin as add-on Treatment in Covid-19 Infected Patients
Brief Title: Escin in Patients With Covid-19 Infection
Acronym: add-on-COV2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: Azienda Ospedaliera Pugliese Ciaccio (Other); Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, Clinical Professor, University of Catanzaro
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: covid-19 add-on therapy
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Coronavirus Infections
MeSH Terms: conditions — Coronavirus Infections | interventions — Escin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- oral escin group (Experimental): Standard therapy+Escin tablet 40mg*3, os for 12 days
  Interventions: Drug: Escin; Drug: standard therapy
- control group (Sham Comparator): standard therapy
  Interventions: Drug: standard therapy
- parenteral escin group (Experimental): standard treatment + sodium Escinate 20mg iv/day for 12 days
  Interventions: Drug: Escin; Drug: standard therapy

INTERVENTIONS:
Drug: Escin — treatment with escin or escinate sodium
  Arms: oral escin group; parenteral escin group
Drug: standard therapy — antiviral drugs

SUMMARY:
In December 2019,a new type of pneumonia caused by the coronavirus (COVID-2019) broke out in Wuhan ,China, and spreads quickly to other Chinese cities and 28 countries. More than 70000 people were infected and over 2000 people died all over the world. There is no specific drug treatment for this disease. Considering that lung damage is related to both viral infection and burst of cytokines, our idea is to evaluate the efficacy and safety of escin as add-on treatment to conventional antiviral drugs in COVID-19 infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years, extremes included, male or female
* Positivity to covid-19 screening test in molecular biology
* In escin group: Low response to standard treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding.
* patients with previous history to allergy
* patients meet the contraindications of escin
* Patients have any condition that in the judgement of the Investigators would make the subject inappropriate for entry into this study.
* patients can't take drugs orally

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | up to 30 days
  All cause mortality
Clinical status evaluated in agreement with guidelines | up to 30 days
  mild type：no No symptoms, Radiological examination: no pneumonia; possible mild increase in C-reactive portein 2, moderate type: fever, cough, or other respiratory symptoms. Radiological examination: pneumonia, SpO2>93% without oxygen inhalation ; increase in C reactive protein, 3: severe type: a. Rate ≥30bpm；b. Pulse Oxygen Saturation (SpO2)≤93% without oxygen inhalation，c. PaO2/FiO2(fraction of inspired oxygen )≤300mmHg ；4. Critically type：match any of the follow: a. need mechanical ventilation; b. shock; c. (multiple organ dysfunction syndrome) MODS

SECONDARY OUTCOMES:
The differences in oxygen intake methods | up to 30 days
  Pulse Oxygen Saturation(SpO2)>93%，1. No need for supplemental oxygenation; 2. nasal catheter oxygen inhalation（oxygen concentration%,The oxygen flow rate：L/min）；3. Mask oxygen inhalation（oxygen concentration%,The oxygen flow rate：L/min）；4. Noninvasive ventilator oxygen supply（Ventilation mode,oxygen concentration%,The oxygen flow rate：L/min,）；5. Invasive ventilator oxygen supply（Ventilation mode,oxygen concentration%,The oxygen flow rate：L/min,）
Time of hospitalization (days) | up to 30 days
  days
Time of hospitalization in intensive care units | up to 30 days
  days
Pulmonary function | up to 3 months after discharge
  forced expiratory volume at one second ,maximum voluntary ventilation at 1month，2month，3month after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Luca Gallelli, Catanzaro, Italy